CLINICAL TRIAL: NCT05909657
Title: Access to Care for SCD Management in Jamaica: Enablers and Barriers to Hydroxyurea Utilization
Brief Title: Enablers and Barriers to Hydroxyurea Use for Sickle Cell Disease Jamaica
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Other Study IDs: CREC-MN.008,2022/2023
Record Dates: First submitted 2023-04-06; First posted 2023-06-18 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
Keywords: hydroxyurea; access to care; Jamaica
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sickle Cell Disease patients = or > 18 years in Jamaica: surveys, interviews
  Interventions: Other: questionnaires (surveys)
- Adult Caregivers of Sickle Cell Disease Children/Adolescents under 18 years: surveys, interviews
  Interventions: Other: questionnaires (surveys)
- Healthcare Providers: SCD Physicians, Nurses and Pharmacists: surveys and interviews
  Interventions: Other: questionnaires (surveys)

INTERVENTIONS:
Other: questionnaires (surveys) — Mixed-methods study. Both the qualitative interview guides and the questionnaire surveys are adapted from the Sickle Cell Disease Implementation Consortium (SCDIC) project which is a multicentre study occurring in the United States.
  Other Names: in-depth interviews

SUMMARY:
Sickle cell disease (SCD) is associated with a lifetime of medical and socio-behavioural complications that require coordination of care from multidisciplinary teams. Access to adequate care for SCD is important as inadequate access can contribute to increased acute care utilization, disjointed care delivery, and earlier mortality for many SCD patients. Hydroxyurea (HU) is the first drug approved for the treatment of SCD and improves many adverse outcomes of SCD and yet its use remains sub-optimal. This mixed-methods study aims to identify the barriers and enablers that SCD patients, caregivers of children (under age 18 years), and health care providers (including physicians, nurses and pharmacists) identify for health care access and HU utilization. The findings may guide development and implementation of strategies to improve access to SCD healthcare and HU uptake which may result in significant benefits to patients, families and the healthcare system including possible reduction in healthcare utilization. Participants will be recruited from the Sickle Cell Unit, Kingston and from all four Jamaican regional health authorities. Questionnaires and interview guides for provider and patient/caregiver assessments are adapted, with permission, from the Sickle Cell Disease Implementation Consortium tools. The study will also examine data on HU usage from the National Health Fund of Jamaica since its addition of SCD to its list of chronic illnesses in 2015. All data collected will be de-identified and maintained in a secure database, with access limited to key personnel. There is minimal risk to participants. Participants will be selected only because of the specific problem under investigation, and not because of easy availability, diminished autonomy, or social bias.

ELIGIBILITY:
Inclusion Criteria:

* SCD Patients (ages 18 and over)
* Adult Caregivers of SCD Children/Adolescents under 18 years
* Healthcare Providers: Physicians, Nurses and Pharmacists who treat and interact with sickle cell patients

Exclusion Criteria:

* SCD patients below age 18 years
* SCD patients who are acutely ill

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruitment Patients and caregivers of children (ages < 18 years) with SCD will be recruited islandwide- specifically from the Sickle Cell Unit (SCU) located at the University of the West Indies (UWI) campus and from all four regional health authorities. Patients will be recruited when in a well state. Similarly healthcare providers - Physicians, Registered Nurses, and Pharmacists- will be recruited from each region. For the desk review there would be interviews conducted with the Director of logistics and the Director of individual benefits - NHF, Policy Director or designee at MOHW, NCD director - MOHW and the Health Service Director - MOHW.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
surveys to determine patient and caregiver access to HU and perceived barriers to HU use for SCD in Jamaica | 18 months
  1. Determine where people living with SCD access care and perceived barriers to receiving care.
  In-depth interview guides will be adapted, with permission from the Sickle Cell Disease Implementation Consortium tools.
in-depth interviews to determine patient and caregiver access to HU and perceived barriers to HU use for SCD in Jamaica | 18 months
  Determine where people living with SCD access care and perceived barriers to receiving care.
  In-depth interview guides will be adapted, with permission from the Sickle Cell Disease Implementation Consortium tools.
surveys to asses patients and caregivers experience using HU for SCD in Jamaica | 18 Months
  3. Assess the acceptability, accessibility, adherence, and satisfaction with HU therapy among patients and caregivers of patients with SCD cross sectional study using questionnaires adapted from the Sickle Cell Disease Implementation Consortium tools will be administered to patients, caregivers and healthcare professionals.
  In-depth interview guides will also be adapted, with permission from the Sickle Cell Disease Implementation Consortium tools, will be used
in-depth interviews to asses patients and caregivers experience using HU for SCD in Jamaica | 18 Months
  Assess the acceptability, accessibility, adherence, and satisfaction with HU therapy among patients and caregivers of patients with SCD cross sectional study using questionnaires adapted from the Sickle Cell Disease Implementation Consortium tools will be administered to patients, caregivers and healthcare professionals. All measures will be self reported to assess acceptability, accessibility, adherence, and satisfaction with HU therapy based on experience and knowledge already held. Lower scores for acceptability, accessibility, adherence, and satisfaction connote a worse outcome, and better outcomes are associated with higher scores for these measures.
  In-depth interview guides will also be adapted, with permission from the Sickle Cell Disease Implementation Consortium tools, will be used
examine healthcare providers knowledge and attitudes toward providing HU for SCD in Jamaica using surveys | 18 months
  5. Assess the knowledge, attitudes and barriers perceived by healthcare providers in provision of HU treatment cross sectional study using questionnaires adapted from the Sickle Cell Disease Implementation Consortium tools will be administered to patients, caregivers and healthcare professionals.
In-depth interviews to examine healthcare providers knowledge and attitudes toward providing HU for SCD in Jamaica | 18 months
  Assess the knowledge, attitudes and barriers perceived by healthcare providers in provision of HU treatment by employing the use of in-depth interview guides adapted, with permission from the Sickle Cell Disease Implementation Consortium tools.
Desk review of supply and benefits used for HU will be conducted in the study with the aim to identify potential gaps in the health care service delivery that may reduce the uptake of hydroxyurea by persons with sickle cell disease | 18 months
  We will describe the process used to keep pharmacy supply of HU sufficient for numbers of patients living with SCD in different areas, how this supply of HU is prescribed to patients, when it is dispensed to patients and from which pharmacies (government or private), and which government or private insurance benefits are used by patients for the purposes of acquiring HU. This information will be collected to examine the efficiency of the health system in supplying HU to the SCD population A desk review will be conducted in the initial stages of the study with the aim to identify potential gaps in the health care service delivery that may reduce the uptake of hydroxyurea by persons with sickle cell disease. This will provide an evaluation of data quality. This information will also be used for internal consistency, external comparisons and external consistency of population data. A guide from the Sickle Cell Disease Implementation Consortium tools, will be used with permission.
A desk review assessment of the cost to patients in the health care system to deliver HU for patients living with Sickle Cell Disease in Jamaica | 10 months
  8. Examine the cost associated with the use of HU in the health system to the SCD population A desk review will be conducted in the initial stages of the study with the aim to identify potential gaps in the health care service delivery that may reduce the uptake of hydroxyurea by persons with sickle cell disease.
  A guide from the Sickle Cell Disease Implementation Consortium tools, will be used with permission.
Assessment of the health care system to deliver HU for patients living with Sickle Cell Disease in Jamaica by doing a desk review and defining where (pharmacies - private, government, or hospital) HU is made available in Jamaica. | 18 months
  9. A count and qualitative examination of the availability of HU within the health system to the SCD population A desk review will be performed in the initial stages of the study with the aim to identify potential gaps in the health care service delivery that may reduce the uptake of hydroxyurea by persons with sickle cell disease specifically if these gaps might include where HU is sourced in Jamaican pharmacies (as these are the last link in delivery of HU to patients with SCD).
  A guide from the Sickle Cell Disease Implementation Consortium tools, will be used with permission.

CONTACTS AND LOCATIONS:
Locations (1):
- Sickle Cell Unit - Caribbean Institute for Health Research, Kingston, Saint Andrew Parish, Jamaica

IPD SHARING:
Plan to Share IPD: No
Patients will be recruited when in a well state. Similarly healthcare providers - Physicians, Registered Nurses, and Pharmacists- will be recruited from each region. Those who choose to participate in the in-depth interviews will be invited to do so face to face or virtually using platforms such as Zoom or WhatsApp. The information obtained via the desk review will be anonymized as much as possible, no names will be utilized in the reporting of the transcripts. All study procedures will be conducted only once informed consent has been obtained.